CLINICAL TRIAL: NCT03170726
Title: Impact of Preemptive Intravenous Ibuprofen on Intraoperative Analgesia in Third Molar Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERZINCAN UNIVERSITY 9
Record Dates: First submitted 2017-05-20; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Preemptive Intravenous Ibuprofen; Intraoperative Analgesia
Keywords: Preemptive intravenous ibuprofen; Intraoperative analgesia; Third molar tooth surgery
MeSH Terms: interventions — dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- arveles (Active Comparator): Ibuprofen 800 mg in normal saline 150 cc and dexketoprofen (50 mg) before operation will be given in 30 minutes
  Interventions: Drug: arveles; Drug: intrafen 800 mg; Other: plasebos
- intrafen (Active Comparator): intrafen 800 mg in normal saline 150 cc before operation will be given in 30 minutes
  Interventions: Drug: arveles; Drug: intrafen 800 mg; Other: plasebos
- plasebos (Placebo Comparator): 150 cc normal saline will be given in 30 minutes during preoperative period
  Interventions: Drug: arveles; Drug: intrafen 800 mg; Other: plasebos

INTERVENTIONS:
Drug: arveles — Intraoperative and postoperative pain values between these three groups will be compared.
  Other Names: dexketoprofen
Drug: intrafen 800 mg — ibuprofen 800 mg in normal saline 150 cc before operation will be given in 30 minutes. Intraoperative and postoperative pain values between these three groups will be compared.
  Other Names: ibuprofen i.v.
Other: plasebos — normal saline 150 cc before operation will be given in 30 minutes. Intraoperative and postoperative pain values between these three groups will be compared.

SUMMARY:
This study was planned to evaluate the analgesic efficacy of preemptive intravenous (iv) ibuprofen on pain occurring during and after the mandibular third molar surgeon

ELIGIBILITY:
Inclusion Criteria:

* Patients who are to be elected third molar tooth extraction
* Patients between the ages of 20-35
* Patients who are symptomatic
* Third molar tooth angular or horizontal settled patients

Exclusion Criteria:

* Patients who refuse to participate in the study
* Patients under 20 years old, over 35 years old
* Patients who are allergic to known non-steroidal anti-inflammatory drugs
* Pregnant patients
* Patients with severe liver failure,
* patients with severe renal insufficiency

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-10-30 (Estimated); Study Completion 2017-11-15 (Estimated)

PRIMARY OUTCOMES:
intraoperative pain as assessed by visual analogue scale | 5 month
  Assessment of Preemptive intravenous ibuprofen on intraoperative analgesic efficacy in 3. molar tooth extraction

SECONDARY OUTCOMES:
postoperative pain as assessed by visual analogue scale | 5 month
  postoperative analgesic contribution of preemptively administered intravenous ibuprofen.

CONTACTS AND LOCATIONS:
Overall Officials: ilke kupeli, Principal Investigator — Erzincan University
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jerjes W, El-Maaytah M, Swinson B, Banu B, Upile T, D'Sa S, Al-Khawalde M, Chaib B, Hopper C. Experience versus complication rate in third molar surgery. Head Face Med. 2006 May 25;2:14. doi: 10.1186/1746-160X-2-14. PMID 16725024
- [Background] Oscier CD, Milner QJ. Peri-operative use of paracetamol. Anaesthesia. 2009 Jan;64(1):65-72. doi: 10.1111/j.1365-2044.2008.05674.x. PMID 19087009
- [Background] Hariharan S, Moseley H, Kumar A, Raju S. The effect of preemptive analgesia in postoperative pain relief--a prospective double-blind randomized study. Pain Med. 2009 Jan;10(1):49-53. doi: 10.1111/j.1526-4637.2008.00547.x. PMID 19222770
- [Result] Trampitsch E, Pipam W, Moertl M, Sadjak A, Dorn C, Sittl R, Likar R. [Preemptive randomized, double-blind study with lornoxicam in gynecological surgery]. Schmerz. 2003 Jan;17(1):4-10. doi: 10.1007/s00482-001-0129-7. German. PMID 12579384
- [Result] Buvanendran A, Kroin JS. Multimodal analgesia for controlling acute postoperative pain. Curr Opin Anaesthesiol. 2009 Oct;22(5):588-93. doi: 10.1097/ACO.0b013e328330373a. PMID 19606021